CLINICAL TRIAL: NCT04884217
Title: Treatment of Dry Eye Disease Using Pro-ocular™ - A Proof of Concept, Safety, and Efficacy Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: PharmaDax Inc. (Industry)
Collaborators: Glia, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DE-2
Record Dates: First submitted 2021-05-10; First posted 2021-05-12 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Dry Eye Syndrome; Keratoconjunctivitis Sicca
Keywords: Dry Eye; Dry Eye Disease; Evaporative Dry Eye; Evaporative Dry Eye Disease; Keratoconjuncitivitis Sicca; Sjogren's Sydrome
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pro-ocular™ (Active Comparator): Pro-ocular™ Topical Gel
  Interventions: Drug: Pro-ocular™ Topical Gel
- Placebo (Placebo Comparator): Placebo Topical Gel
  Interventions: Drug: Placebo Topical Gel

INTERVENTIONS:
Drug: Pro-ocular™ Topical Gel — Pro-ocular™ Topical Gel 1% is applied dermally to the forehead twice-daily
  Other Names: PG101
  Arms: Pro-ocular™
Drug: Placebo Topical Gel — Placebo is a toopical gel without active ingredient applied dermally to the forehead twice-daily
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of 1% Pro-ocular topical gel administered twice daily for 12 weeks in treatment of Dry Eye Disease

DETAILED DESCRIPTION:
Pro-ocular™ 1% topical gel his demonstrated efficacy in rapidly reducing or eliminating dry eye symptoms, and after multiple doses, the signs and symptoms of ocular surface disease including dry eye disease.

Study DE-2 is single center, randomized, double-masked, placebo-controlled, parallel-group study designed to evaluate the safety and efficacy of 1% Pro-ocular topical gel administered twice daily for 12 weeks for treatment of Dry Eye Disease. The approximately 80 subjects will be randomized 1:1, active drug:placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of any race, at least 20 years of age at Visit 1 Screening.
2. Has a subject reported history (including physician diagnosis) of dry eye disease in both eyes for at least 3 months prior to Visit 1.
3. Has SANDE score ≥50 in either frequency or severity of symptoms of dryness and/or irritation at Visit 1.
4. Have all of the following in the same eye at Visit 1:

   1. Fluorescein Tear Break-Up Time of ≤5 seconds.
   2. Corneal fluorescein staining score of moderate or more in any field (inferior, superior or central).
   3. Report a severity score of moderate or more on ocular dryness and at least one of the other symptoms on the GLIA Ocular Surface Disease Symptoms Questionnaire.
5. Has provided written informed consent.
6. Be able and willing to follow oral and written instructions, including participation in all study assessments and visits.

Exclusion Criteria:

1. Comorbidity with other severe or chronic eye conditions that in the judgment of the investigator will interfere with study assessments, such as but not limited to corneal opacities and scars, dystrophies, epithelial scarring, infections, history of blood clots, etc.
2. Has infections, or inflammatory skin lesion in or around the dosing area.
3. Best corrected visual acuity baseline <20/200.
4. Has a condition or history that, in the opinion of the investigator, may interfere significantly with the subject's participation in the study.
5. Wear contact lens within 7 days prior to Visit 1.
6. Anticipate change of vision correction or anticipate any ocular procedures during study period.
7. A woman who is pregnant or testing positive in the blood pregnancy test at screening, nursing an infant, or planning a pregnancy.
8. Has a known adverse reaction and/or sensitivity to the study drug or its components.
9. Use of topical ocular cyclosporine (e.g. Restasis®), lifitegrast (Xiidra®), diquafosol (Diquas®), eye gels, eye ointments, any administration route of steroids, anti-histamines, antipsychotics, antidepressants and NSAIDs within 30 days prior to Visit 1.
10. Routine use (more than once a week) of a chlorinated swimming pool during study period.
11. Unwilling or unable to cease using the following medications during the study period (from Visit 1 to Visit 6): Topical ocular cyclosporine (e.g. Restasis®), lifitegrast (Xiidra®), diquafosol (Diquas®), eye gels, eye ointments, any administration route of steroids, anti-histamines, antipsychotics, antidepressants and NSAIDs..
12. Unwilling to cease the use of sunscreen and face scrubs on the forehead or eye area during study period.
13. Smoke within 3 months prior to Visit 1.
14. Ongoing glaucoma treatment within 30 days prior to Visit 1 and during study period.
15. Currently enrolled in an investigational drug or device study within 30 days prior to Visit 1 and during study period.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-05-20 (Estimated); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in SANDE (Symptom Assessment iN Dry Eye) Questionnaire Frequency score | 2 weeks
  Change from baseline in SANDE symptoms frequency score (0-100 worst)
Change in corneal (central) fluorescein staining score | 4 weeks
  Change from baseline in score on a visual analog scale (0-10 worst)

SECONDARY OUTCOMES:
Change in SANDE (Symptom Assessment iN Dry Eye) Questionnaire Global score | 2 weeks
  Change from baseline in SANDE symptoms global score (0-100 worst)
Change in SANDE (Symptom Assessment iN Dry Eye) Questionnaire Global score | 4 weeks
  Change from baseline in SANDE symptoms global score (0-100 worst)
Change in SANDE (Symptom Assessment iN Dry Eye) Questionnaire Global score | 8 weeks
  Change from baseline in SANDE symptoms global score (0-100 worst)
Change in SANDE (Symptom Assessment iN Dry Eye) Questionnaire Global score | 12 weeks
  Change from baseline in SANDE symptoms global score (0-100 worst)
Change in SANDE (Symptom Assessment iN Dry Eye) Questionnaire Frequency score | 4 weeks
  Change from baseline in SANDE symptoms frequency score (0-100 worst)
Change in SANDE (Symptom Assessment iN Dry Eye) Questionnaire Frequency score | 8 weeks
  Change from baseline in SANDE symptoms frequency score (0-100 worst)
Change in SANDE (Symptom Assessment iN Dry Eye) Questionnaire Frequency score | 12 weeks
  Change from baseline in SANDE symptoms frequency score (0-100 worst)
Change in SANDE (Symptom Assessment iN Dry Eye) Questionnaire Severity score | 2 weeks
  Change from baseline in SANDE symptoms severity score (0-100 worst)
Change in SANDE (Symptom Assessment iN Dry Eye) Questionnaire Severity score | 4 weeks
  Change from baseline in SANDE symptoms severity score (0-100 worst)
Change in SANDE (Symptom Assessment iN Dry Eye) Questionnaire Severity score | 8 weeks
  Change from baseline in SANDE symptoms severity score (0-100 worst)
Change in SANDE (Symptom Assessment iN Dry Eye) Questionnaire Severity score | 12 weeks
  Change from baseline in SANDE symptoms severity score (0-100 worst)
Change in GLIA (Ocular Surface Disease Symptoms Questionnaire) ocular discomfort score | 1 hour
  Change from baseline in GLIA OSDSQ ocular discomfort score (0-10 worst)
Change in GLIA (Ocular Surface Disease Symptoms Questionnaire) ocular discomfort score | 2 weeks
  Change from baseline in GLIA OSDSQ ocular discomfort score (0-10 worst)
Change in GLIA (Ocular Surface Disease Symptoms Questionnaire) ocular discomfort score | 4 weeks
  Change from baseline in GLIA OSDSQ ocular discomfort score (0-10 worst)
Change in GLIA (Ocular Surface Disease Symptoms Questionnaire) ocular discomfort score | 8 weeks
  Change from baseline in GLIA OSDSQ ocular discomfort score (0-10 worst)
Change in GLIA (Ocular Surface Disease Symptoms Questionnaire) ocular discomfort score | 12 weeks
  Change from baseline in GLIA OSDSQ ocular discomfort score (0-10 worst)
Change in GLIA (Ocular Surface Disease Symptoms Questionnaire) sum of scores | 1 hour
  Change from baseline in GLIA OSDSQ sum of scores (highest worst)
Change in GLIA (Ocular Surface Disease Symptoms Questionnaire) sum of scores | 2 weeks
  Change from baseline in GLIA OSDSQ sum of scores (highest worst)
Change in GLIA (Ocular Surface Disease Symptoms Questionnaire) sum of scores | 4 weeks
  Change from baseline in GLIA OSDSQ sum of scores (highest worst)
Change in GLIA (Ocular Surface Disease Symptoms Questionnaire) sum of scores | 8 weeks
  Change from baseline in GLIA OSDSQ sum of scores (highest worst)
Change in GLIA (Ocular Surface Disease Symptoms Questionnaire) sum of scores | 12 weeks
  Change from baseline in GLIA OSDSQ sum of scores (highest worst)
Change in Tear Film Grading by TearScan examination | 1 hour
  Change from baseline in tear film grade (0-3 best)
Change in Tear Film Grading by TearScan examination | 2 weeks
  Change from baseline in tear film grade (0-3 best)
Change in Tear Film Grading by TearScan examination | 4 weeks
  Change from baseline in tear film grade (0-3 best)
Change in Tear Film Grading by TearScan examination | 8 weeks
  Change from baseline in tear film grade (0-3 best)
Change in Tear Film Grading by TearScan examination | 12 weeks
  Change from baseline in tear film grade (0-3 best)
Change in Meibography score by Keratograph® | 12 weeks
  Change from baseline using Grades 0 to 3 (0 no loss to 3 >2/3 loss)
Change in Tear Meniscus Height (TMH) by Keratograph® | 1 hour
  Change from baseline in mm TMH (higher is better)
Change in Tear Meniscus Height (TMH) by Keratograph® | 4 weeks
  Change from baseline in mm TMH (higher is better)
Change in Tear Meniscus Height (TMH) by Keratograph® | 8 weeks
  Change from baseline in mm TMH (higher is better)
Change in Tear Meniscus Height (TMH) by Keratograph® | 12 weeks
  Change from baseline in mm TMH (higher is better)
Change in Non-Invasive Keratograph® Tear Break-Up Time (NIKBUT) | 1 hour
  Change from baseline in NIKBUT in seconds (longer is better)
Change in Non-Invasive Keratograph® Tear Break-Up Time (NIKBUT) | 4 weeks
  Change from baseline in NIKBUT in seconds (longer is better)
Change in Non-Invasive Keratograph® Tear Break-Up Time (NIKBUT) | 8 weeks
  Change from baseline in NIKBUT in seconds (longer is better)
Change in Non-Invasive Keratograph® Tear Break-Up Time (NIKBUT) | 12 weeks
  Change from baseline in NIKBUT in seconds (longer is better)
Change in Bulbar redness score by Keratograph® | 1 hour
  Change from baseline in Bulbar redness score (highest is worst)
Change in Bulbar redness score by Keratograph® | 4 weeks
  Change from baseline in Bulbar redness score (highest is worst)
Change in Bulbar redness score by Keratograph® | 8 weeks
  Change from baseline in Bulbar redness score (highest is worst)
Change in Bulbar redness score by Keratograph® | 12 weeks
  Change from baseline in Bulbar redness score (highest is worst)
Change in tear film osmolarity by TearLab™ osmolarity system | 1 hour
  Change from baseline in mOsms/L (higher value is worse)
Change in tear film osmolarity by TearLab™ osmolarity system | 2 weeks
  Change from baseline in mOsms/L (higher value is less sensitive)
Change in corneal sensitivity using Cochet-Bonnet esthesiometer | 1 hour
  Change from baseline in mm Hg (higher is less sensitive)
Change in corneal sensitivity using Cochet-Bonnet esthesiometer | 2 weeks
  Change from baseline in mm Hg (higher is less sensitive)
Change in corneal sensitivity using Cochet-Bonnet esthesiometer | 4 weeks
  Change from baseline in mm Hg (higher is less sensitive)
Change in corneal sensitivity using Cochet-Bonnet esthesiometer | 8 weeks
  Change from baseline in mm Hg (higher is less sensitive)
Change in corneal sensitivity using Cochet-Bonnet esthesiometer | 12 weeks
  Change from baseline in mm Hg (higher is less sensitive)
Change in Fluorescein Tear Break-Up Time (FBUT) | 1 hour
  Change from baseline in FBUT in seconds (longer is better)
Change in Fluorescein Tear Break-Up Time (FBUT) | 4 weeks
  Change from baseline in FBUT in seconds (longer is better)
Change in Fluorescein Tear Break-Up Time (FBUT) | 8 weeks
  Change from baseline in FBUT in seconds (longer is better)
Change in Fluorescein Tear Break-Up Time (FBUT) | 12 weeks
  Change from baseline in FBUT in seconds (longer is better)
Change in corneal (central) fluorescein staining score | 2 weeks
  Change from baseline in central corneal fluorescein staining score (0-10 worst)
Change in corneal (central) fluorescein staining score | 8 weeks
  Change from baseline in central corneal fluorescein staining score (0-10 worst)
Change in corneal (central) fluorescein staining score | 12 weeks
  Change from baseline in central corneal fluorescein staining score (0-10 worst)
Change in corneal (inferior) fluorescein staining score | 2 weeks
  Change from baseline in inferior corneal fluorescein staining score (0-10 worst)
Change in corneal (inferior) fluorescein staining score | 4 weeks
  Change from baseline in inferior corneal fluorescein staining score (0-10 worst)
Change in corneal (inferior) fluorescein staining score | 8 weeks
  Change from baseline in inferior corneal fluorescein staining score (0-10 worst)
Change in corneal (inferior) fluorescein staining score | 12 weeks
  Change from baseline in inferior corneal fluorescein staining score (0-10 worst)
Change in corneal (superior) fluorescein staining score | 2 weeks
  Change from baseline in superior corneal fluorescein staining score (0-10 worst)
Change in corneal (superior) fluorescein staining score | 4 weeks
  Change from baseline in superior corneal fluorescein staining score (0-10 worst)
Change in corneal (superior) fluorescein staining score | 8 weeks
  Change from baseline in superior corneal fluorescein staining score (0-10 worst)
Change in corneal (superior) fluorescein staining score | 12 weeks
  Change from baseline in superior corneal fluorescein staining score (0-10 worst)
Change in corneal fluorescein staining sum of scores | 2 weeks
  Change from baseline in corneal fluorescein staining sum of scores (0-30 worst)
Change in corneal fluorescein staining sum of scores | 4 weeks
  Change from baseline in corneal fluorescein staining sum of scores (0-30 worst)
Change in corneal fluorescein staining sum of scores | 8 weeks
  Change from baseline in corneal fluorescein staining sum of scores (0-30 worst)
Change in corneal fluorescein staining sum of scores | 12 weeks
  Change from baseline in corneal fluorescein staining sum of scores (0-30 worst)
Change in conjunctival fluorescein staining sum of scores | 2 weeks
  Change from baseline in conjunctival fluorescein staining sum of scores (0-30 worst)
Change in conjunctival fluorescein staining sum of scores | 4 weeks
  Change from baseline in conjunctival fluorescein staining sum of scores (0-30 worst)
Change in conjunctival fluorescein staining sum of scores | 8 weeks
  Change from baseline in conjunctival fluorescein staining sum of scores (0-30 worst)
Change in conjunctival fluorescein staining sum of scores | 12 weeks
  Change from baseline in conjunctival fluorescein staining sum of scores (0-30 worst)
Change in lissamine green staining (corneal and conjunctival) sum of scores | 2 weeks
  Change from baseline in lissamine green staining (corneal and conjunctival) sum of scores
Change in lissamine green staining (corneal and conjunctival) sum of scores | 4 weeks
  Change from baseline in lissamine green staining (corneal and conjunctival) sum of scores (higher is worse)
Change in lissamine green staining (corneal and conjunctival) sum of scores | 8 weeks
  Change from baseline in lissamine green staining (corneal and conjunctival) sum of scores (higher is worse)
Change in lissamine green staining (corneal and conjunctival) sum of scores | 12 weeks
  Change from baseline in lissamine green staining (corneal and conjunctival) sum of scores (higher is worse)
Change in conjunctival hyperemia (by slit lamp biomicroscopy) | 2 weeks
  Change from baseline in conjunctival hyperemia score (0-10 worst)
Change in conjunctival hyperemia (by slit lamp biomicroscopy) | 4 weeks
  Change from baseline in conjunctival hyperemia score (0-10 worst)
Change in conjunctival hyperemia (by slit lamp biomicroscopy) | 8 weeks
  Change from baseline in conjunctival hyperemia score (0-10 worst)
Change in conjunctival hyperemia (by slit lamp biomicroscopy) | 12 weeks
  Change from baseline in conjunctival hyperemia score (0-10 worst)

CONTACTS AND LOCATIONS:
Overall Officials: Peichun Kuo, Study Director — PharmaDax Inc.
Locations (1):
- Tri-Service General Hospital, National Defense Medical Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No